CLINICAL TRIAL: NCT01436695
Title: Safety and Feasibility of Using Epicall for Monitoring Pre-seizure Biomarkers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Epicall LTD (Industry)
Responsible Party: Sponsor
Other Study IDs: EPC - 01
Record Dates: First submitted 2011-09-17; First posted 2011-09-20 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2011-09

CONDITIONS: Seizure
Keywords: seizure early detection
MeSH Terms: conditions — Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Epicall group: patients will be connected to Epicall sensor
  Interventions: Device: Epicall

INTERVENTIONS:
Device: Epicall — The Epicall system is intended for early detection of seizure by monitoring pre-seizure biomarkers.

SUMMARY:
Epilepsy is a syndrome of episodic brain dysfunction characterized by recurrent seemingly unpredictable spontaneous seizures. The occurrence of the seizure in patients without any forewarning is the most debilitating aspect of the disease.

The Epicall system is intended for early detection of seizure related life threatening events by monitoring per-seizures biomarkers. The system is based on a sticker placed on the side of the face. The external sticker incorporates EOG (electrooculograph electrode) and PPG (photoplethysmograph electrode) sensors for continuous monitoring of:

1. Heart Rate (base line, increase, decrease, asystole).
2. Extra ocular eye movement (blinking, eye deviation, roving eye movements).

ELIGIBILITY:
Inclusion Criteria:

* Children age 1 year -18 years old.
* Hospitalized patient who is diagnosed with epilepsy.
* Patient's parents/care giver able to comprehend and give informed consent for participation in this study.
* Patient's parents/care giver must commit to both screening and monitoring visits.
* Patient's parents/care giver must sign the Informed Consent Form.

Exclusion Criteria:

* Patient with any infection / abscess / bleeding / blister / crack / edema / fissure / ulcer / pain in monitoring electrode area
* General weakness.
* Patient's parents/care giver objects to the study protocol.
* Concurrent participation in any other clinical study.
* Physician objection.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Hospitalized patients who diagnosed with epilepsy and meet all of the eligibility criteria will be recruited for the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Lack of adverse events | 1-2 weeks

SECONDARY OUTCOMES:
Epicall feasibility for monitoring pre-seizure biomarkers | 1-2 weeks
  Feasibility of using the Epicall for monitoring pre-seizure biomarkers will be established by the correlation between Epicall and ECG heart rate measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Eli Heyman, Dr, Principal Investigator — Asaf-Harofeh Medical Center, Zrifin Israel
Locations (1):
- Asaf Harofeh Medical Center, Zrifin, Israel